CLINICAL TRIAL: NCT04899414
Title: Study Evaluating the Safety and Efficacy of the Dexamethasone, Azacytidine, Pegaspargase, Tislelizumab With NK/T Cell Lymphoma
Brief Title: Dexamethasone, Azacytidine,Pegaspargase and Tislelizumab for NK/T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Zhu, Dr., Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAPT for NKTCL
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: NK/T Cell Lymphoma
Keywords: DAPT; Tislelizumab; Non- upper aerodigestive tract NK/T- cell lymphoma; R/R NK/T- cell lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Dexamethasone; Azacitidine; pegaspargase; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stage III/IV or Stage I/II NUAT- NKTCL or Relapsed or Refractory NK/T- cell lymphoma (Experimental): 4-6 cycles of induction DAPT followed by Auto HSCT as consolidation for CR/PR fit patients ,then by PD-1 as maintenance treatment (up to 16 cycles) for received Auto-HSCT
  Interventions: Drug: Dexamethasone, azacytidine, Pegaspargase, Tislelizumab

INTERVENTIONS:
Drug: Dexamethasone, azacytidine, Pegaspargase, Tislelizumab — Dexamethasone 40mg intravenously daily on day 1-4; azacytidine 100mg intravenously daily on day 1-5; Pegaspargase 3750 IU intravenously daily on day 1； Tislelizumab 200 mg IV on Day 1 of each 21-day as a cycle.

SUMMARY:
The optimal first-line treatment for extra-nodal NK/T-cell lymphoma (ENKTL) has not been well-defined. This phase II study aimed to evaluate the efficacy and safety of Dexamethasone, azacytidine, Pegaspargase, Tislelizumab (DAPT) regimen for patients with newly diagnosed advanced stage ENKTL

, non-upper aerodigestive tract NK/T- cell lymphoma（NUAT- NKTCL）and relapsed refractory NK/T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years ,Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* patients with confirmed pathological diagnosis of ENKTL as defined by WHO criteria
* at least one measurable lesion
* hemoglobin ≥90 g/l, absolute neutrophil count ≥ 1.5 × 10^9/L, platelets ≥ 75 ×10^9/L), ALT≤ 2 times upper limit of normal, serum creatinine ≤1.5 times upper limit of normal （If the above indicators are abnormal but are caused by the primary disease as assessed by the clinician, the treatment can be enrolled according to the clinical actual situation）
* There was no other serious disease in conflict with this program
* Adequate respiratory function
* Adequate bone marrow function
* Adequate renal and hepatic function
* Not pregnant or nursing ,negative pregnancy test
* No other active malignancy requiring therapy
* No other serious or life-threatening condition deemed unacceptable by the principal investigator
* Life expectancy ≥ 3 months
* Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

* NK/T cell lymphoma without confirmed pathological diagnosis;
* Patients with early stage upper aerodigestive tract NK/T- cell lymphoma ;
* Patients with drug allergies or metabolic disorders in the program;
* Any uncontrolled medical diseases (including uncontrolled diabetes, severe heart, lung, liver and kidney dysfunction);
* Severe infection (excluding the following: HBsAg or anti-HBc positive patients taking entecavir, tenofovir and other drugs;HCV RNA positive but taking direct anti-HCV drugs);
* Invasion of primary or secondary central nervous system tumor invasion;
* Contradictions to chemotherapy or radiotherapy;
* Previously other malignancy requiring therapy;
* Peripheral nervous system disorder or mental disorder;
* Incapacity for legal conduct, medical or ethical reasons that affect the continuation of the research;
* Other clinical investigators;
* Combination of anti-tumor drugs outside the research program;
* Participants evaluated inappropriate to participate in this study by principal investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-18 (Estimated); Primary Completion 2023-05-18 (Estimated); Study Completion 2023-10-18 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 1-year
  To evaluate the overall response rate of DAPT in the treatment of NK/T cell lymphoma

SECONDARY OUTCOMES:
Complete response rate | 1-year
Progression-free survival | 2-year
Overall survival | 2-year
Adverse events | 1-year

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - National Cancer Center/Cancer Hosptial, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No